CLINICAL TRIAL: NCT03732638
Title: A Phase 2/3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rimegepant in Migraine Prevention
Brief Title: Efficacy and Safety Trial of Rimegepant for Migraine Prevention in Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BHV3000-305
Record Dates: First submitted 2018-11-05; First posted 2018-11-06 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2022-12

CONDITIONS: Migraine
Keywords: Migraine; Prevention; Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DBT Rimegepant/OL Rimegepant (Experimental): DBT Phase (Weeks 1 through 12): Participants received a single oral dose of rimegepant 75 mg tablet every other day (EOD) for 12 weeks.
  OLE Phase (Weeks 13 through 64): Participants who continued to meet study entry criteria and had acceptable laboratory test results per protocol, entered the OLE phase and received a single oral dose of rimegepant 75 mg tablet EOD for 52 weeks. If participants had a migraine on a day that they were not scheduled to dose with rimegepant, they could take one tablet of rimegepant 75 mg on that calendar day to treat a migraine (as needed [PRN] dosing).
  After completing the OLE phase, participants had follow-up safety visits 2 and 8 weeks after the End-of-Treatment (EOT) visit. Participants who did not complete the DBT phase and/or did not enter or complete the OLE phase were to complete the EOT visit, the 2-week follow-up safety visit, and the 8-week follow-up safety visit after their early discontinuation.
  Interventions: Drug: Rimegepant
- DBT Placebo/OL Rimegepant (Placebo Comparator): DBT Phase (Weeks 1 through 12): Participants received a single oral dose of placebo matching to rimegepant tablet EOD for 12 weeks.
  OLE Phase (Weeks 13 through 64): Participants who continued to meet study entry criteria and had acceptable laboratory test results per protocol, entered the OLE phase and received a single oral dose of rimegepant 75 mg tablet EOD for 52 weeks. If participants had a migraine on a day that they were not scheduled to dose with rimegepant, they could take one tablet of rimegepant 75 mg on that calendar day to treat a migraine (PRN dosing).
  After completing the OLE phase, participants had follow-up safety visits 2 and 8 weeks after the End-of-Treatment (EOT) visit. Participants who did not complete the DBT phase and/or did not enter or complete the OLE phase were to complete the EOT visit, the 2-week follow-up safety visit, and the 8-week follow-up safety visit after their early discontinuation.
  Interventions: Drug: Rimegepant; Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75 mg tablet EOD
  Other Names: BHV-3000
Drug: Placebo — Placebo tablet to match rimegepant tablet EOD
  Arms: DBT Placebo/OL Rimegepant

SUMMARY:
The purpose of this is study is to compare the efficacy of BHV-3000 (rimegepant) to placebo as a preventive treatment for migraine, as measured by the reduction in the number of migraine days per month.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least 1 year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, including the following:

   1. Age of onset of migraines prior to 50 years of age
   2. Migraine attacks, on average, lasting 4 - 72 hours if untreated
   3. Per subject report, 4 - 18 migraine attacks of moderate to severe intensity per month within the last 3 months prior to the Screening Visit
   4. 6 or more migraine days during the Observation Period
   5. Not more than 18 headache days during the Observation Period
   6. Ability to distinguish migraine attacks from tension/cluster headaches
   7. Subjects on prophylactic migraine medication are permitted to remain on 1 medication with possible migraine-prophylactic effects if the dose has been stable for at least 3 months prior to the Screening Visit, and the dose is not expected to change during the course of the study.

   Exclusion Criteria:
2. Subject with a history of HIV disease
3. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening
4. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for at least 3 months prior to screening).
5. Subjects with major depressive episode within the last 12 months, major depressive disorder or any anxiety disorder requiring more than 1 medication for each disorder. Medications to treat major depressive disorder or an anxiety disorder must have been at a stable dose for at least 3 months prior to the Screening visit.
6. Subjects with other pain syndromes, psychiatric conditions, dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments
7. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has disease that causes malabsorption
8. Body mass index ≥ 33 kg/m2
9. Subject has current diagnosis of major depressive disorder requiring treatment with atypical antipsychotics, schizophrenia, bipolar disorder, or borderline personality disorder
10. History of gallstones or cholecystectomy.
11. The subject has a history or current evidence of any unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known or suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1590 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (93):
  - MDFirst Research-Chandler, Chandler, Arizona
  - MedPharmics, LLC, Phoenix, Arizona
  - Tucson Neuroscience Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Axiom Research, LLC, Apple Valley, California
  - Axiom Research, LLC, Colton, California
  - eStudySite, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Neurological Research Institute, Santa Monica, California
  - California Neuroscience Research Medical Group, Sherman Oaks, California
  - Ki Health Partners, LLC, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Riverside Clinical Research, Edgewater, Florida
  - Galiz Research, Hialeah, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Qps Mra, Llc, Miami, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - JSV Clinical Research Study Inc., Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Northwest Clinical Trials, Inc, Boise, Idaho
  - R&R Clinical Research, Idaho Falls, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Family Medicine Specialists/CIS, Wauconda, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Heartland Research Associates, LLC, Newton, Kansas
  - Phoenix Medical Research, Prairie Village, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Regeneris Medical, North Attleboro, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Michigan Pain Consultants, Grand Rapids, Michigan
  - MedPharmics, LLC, Biloxi, Mississippi
  - Clinical Research Professionals, Inc., Chesterfield, Missouri
  - StudyMetrix Research, City of Saint Peters, Missouri
  - The Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Nevada Headache Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Central New York Clinical Research, Manlius, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Island Neurological, A Division of Prohealth Care Associates, LLP, Plainview, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - PharmQuest, LLC, Greensboro, North Carolina
  - PMG Research, Raleigh, North Carolina
  - Carolina Research Institute Center, Inc., Shelby, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Hometown Urgent Care, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Neurology Diagnostics Research, Dayton, Ohio
  - Aventiv Research, Inc, Dublin, Ohio
  - Oklahoma Headache Center, Norman, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - BTC of Lincoln, LLC, Lincoln, Rhode Island
  - OnSite Clinical Solutions, Dillon, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Volunteer Research Group, Knoxville, Tennessee
  - Tekton Research, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - North Texas Institute of Neurology & Headache, Frisco, Texas
  - Victorium Clinical Research, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - FMC Science, Lampasas, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - MedStar Georgetown Headache - Georgetown University, McLean, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Women's, Seattle, Washington
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin

REFERENCES:
- [Derived] Kudrow D, Croop RS, Thiry A, Lipton RB. A 52-week open-label extension study to evaluate the safety and efficacy of oral rimegepant for the preventive treatment of migraine. Headache. 2025 Jun 30. doi: 10.1111/head.15002. Online ahead of print. PMID 40583813
- [Derived] Mahon R, Tiwari S, Koch M, Ferraris M, Betts KA, Wang Y, Gao S, Proot P. Comparative effectiveness of erenumab versus rimegepant for migraine prevention using matching-adjusted indirect comparison. J Comp Eff Res. 2024 Mar;13(3):e230122. doi: 10.57264/cer-2023-0122. Epub 2024 Jan 4. PMID 38174577
- [Derived] Powell LC, L'Italien G, Popoff E, Johnston K, O'Sullivan F, Harris L, Croop R, Coric V, Lipton RB. Health State Utility Mapping of Rimegepant for the Preventive Treatment of Migraine: Double-Blind Treatment Phase and Open Label Extension (BHV3000-305). Adv Ther. 2023 Feb;40(2):585-600. doi: 10.1007/s12325-022-02369-x. Epub 2022 Nov 22. PMID 36417057
- [Derived] Croop R, Lipton RB, Kudrow D, Stock DA, Kamen L, Conway CM, Stock EG, Coric V, Goadsby PJ. Oral rimegepant for preventive treatment of migraine: a phase 2/3, randomised, double-blind, placebo-controlled trial. Lancet. 2021 Jan 2;397(10268):51-60. doi: 10.1016/S0140-6736(20)32544-7. Epub 2020 Dec 15. PMID 33338437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 92 sites in the United States.
Pre-assignment Details: A total of 1590 participants were enrolled in the study, of which 747 participants were randomized and 844 were not randomized. Of 747 randomized participants, 741 participants received treatment with blinded study medication. The study was divided into 4 phases: a 4-week observation period (OP), a 12-week double-blind treatment (DBT) phase, a 52-week open-label extension (OLE) phase, and an 8-week follow-up safety phase.
Period: DBT Phase (Weeks 1 to 12)
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Started | 370 | 371
Completed | 316 | 310
Not Completed | 54 | 61
Not completed — Adverse Event | 5 | 2
Not completed — Eligibility failure due to baseline laboratory values | 8 | 13
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 19 | 12
Not completed — Non-compliance | 6 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Protocol deviation | 4 | 5
Not completed — Withdrawal by Subject | 11 | 22
Period: OLE Phase (Weeks 13 to 64)
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Started | 302 (Participants who completed DBT phase and entered the OLE phase) | 301 (Participants who completed DBT phase and entered the OLE phase)
Completed | 209 | 219
Not Completed | 93 | 82
Not completed — Adverse Event | 10 | 9
Not completed — Death | 1 | 1
Not completed — Extension phase eligibility failure due to week 12 laboratory values | 2 | 0
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 19 | 13
Not completed — Non-compliance | 15 | 14
Not completed — Physician Decision | 9 | 9
Not completed — Pregnancy | 2 | 2
Not completed — Protocol deviation | 2 | 3
Not completed — Sponsor Recommendation | 1 | 0
Not completed — Withdrawal by Subject | 29 | 28
Not completed — Other than specified | 1 | 1
Period: Follow-up Phase (up to 72 Weeks)
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Started | 332 (Participants who entered follow-up phase either directly from DBT phase or after OLE phase) | 336 (Participants who entered follow-up phase either directly from DBT phase or after OLE phase)
Completed | 267 | 274
Not Completed | 65 | 62
Not completed — Not reported | 49 | 48
Not completed — Lost to Follow-up | 10 | 6
Not completed — Non-compliance | 2 | 1
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Rimegepant - Randomization Phase: Participants received a single oral dose of rimegepant 75 mg tablet EOD for 12 weeks.
- Placebo - Randomization Phase: Participants received a single oral dose of matching placebo tablet EOD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase | Total
Number analyzed (Participants) | 370 | 371 | 741
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (13.01) | 41.1 (13.13) | 41.2 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 313 | 613
  Male | 70 | 58 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 98 | 203
  Not Hispanic or Latino | 265 | 273 | 538
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 7
  Asian | 1 | 7 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 62 | 49 | 111
  White | 295 | 309 | 604
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Number of Total Migraine Days Per Month in the Last 4 Weeks of the DBT Phase
Description: A migraine day: any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache: a migraine with or without aura, lasting for ≥30 minutes, and meeting at least 1 of the following criteria (a and/or b): a) ≥2 of the following: unilateral location, pulsating quality, moderate to severe pain intensity, aggravation by or causing avoidance of routine physical activity; b) ≥1 of the following: nausea and/or vomiting, photophobia, and phonophobia. If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms.
  Months were defined as 28-day intervals. The change from baseline was calculated as the number of monthly migraine days during the last 4 weeks of the DBT phase (Weeks 9 to 12) minus number of monthly migraine days during the OP.
Time Frame: OP and Weeks 9 to 12 of the DBT phase
Population: The analysis was performed on evaluable modified intent to treat (mITT) participants. Evaluable participants are those with ≥ 14 days of electronic diary efficacy data (not necessarily consecutive) in both the OP and ≥ 1 month (4-week interval) in the DBT phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Total Migraine Days per Month
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 348 | 347
Total Migraine Days per Month | -4.3 [-4.83 to -3.87] | -3.5 [-4 to -3.04]
Statistical Analysis 1: Comparison: Rimegepant - Randomization Phase vs Placebo - Randomization Phase; Test type: Superiority; p = 0.0099, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.46 to -0.20]

2. Secondary Outcome: Number of Participants Who Had ≥ 50% Reduction in Moderate or Severe Migraine Days Per Month in the Last 4 Weeks of the DBT Phase
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (as previously described). If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms. A moderate or severe migraine day was a migraine day of moderate or severe pain intensity. Months were defined as 28-day intervals.
  A reduction of at least 50% in the mean number of moderate or severe monthly migraine days was determined if the number of moderate or severe monthly migraine days in the last 4 weeks of the DBT (Weeks 9 to 12) was less than or equal to half (50%) of the number of moderate or severe monthly migraine days in the OP.
Time Frame: OP and Weeks 9 to 12 of the DBT phase
Population: The analysis was performed on evaluable mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 348 | 347
percentage of participants | 49.1 [43.9 to 54.3] | 41.5 [36.3 to 46.7]
Statistical Analysis 1: Comparison: Rimegepant - Randomization Phase vs Placebo - Randomization Phase; Test type: Superiority; p = 0.0438, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.6, 95% CI 2-sided [0.2 to 14.9]

3. Secondary Outcome: Change From Baseline in the Mean Number of Migraine Days Per Month Over the Entire Course of the DBT Phase
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (as previously described). If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms. Months were defined as 28-day intervals.
  The change from baseline was calculated as the number of monthly migraine days during the DBT phase (Weeks 1 to 12) minus the number of monthly migraine days during the OP.
Time Frame: OP and Weeks 1 to 12 of the DBT phase
Population: The analysis was performed on evaluable mITT participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Total Migraine Days per Month
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 348 | 347
Total Migraine Days per Month | -3.6 [-3.97 to -3.17] | -2.7 [-3.14 to -2.34]
Statistical Analysis 1: Comparison: Rimegepant - Randomization Phase vs Placebo - Randomization Phase; Test type: Superiority; p = 0.0017, Mixed Models Analysis; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.34 to -0.31]

4. Secondary Outcome: Frequency of Use of Rescue Medication Days Per Month in the Last Month of the DBT Phase
Description: A rescue medication day was a day on which the participant took triptan, ergotamine, or other permitted medication to acutely treat headache or aura. Months were defined as 28-day intervals.
Time Frame: Weeks 9 to 12 of the DBT phase
Population: The analysis was performed on evaluable mITT participants
Measure: Least Squares Mean (95% Confidence Interval); unit: rescue medication Days per Month
Groups:
- Placebo - Randomization Phase: Participants received a single oral dose of matching placebo table EOD for 12 weeks.
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 348 | 347
rescue medication Days per Month | 3.7 [3.29 to 4.15] | 4.0 [3.53 to 4.39]
Statistical Analysis 1: Comparison: Rimegepant - Randomization Phase vs Placebo - Randomization Phase; Test type: Superiority; p = 0.3868, Mixed Models Analysis — P-value ≥ 0.05; therefore, all secondary endpoints listed after this endpoint in the hierarchy were not tested; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.80 to 0.31]

5. Secondary Outcome: Change From Baseline in the Mean Number of Total Migraine Days Per Month in the First Month of the DBT Phase
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (as previously described). If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms. Months were defined as 28-day intervals.
  The change from baseline was calculated as the number of monthly migraine days during the first 4 weeks of the DBT phase (Weeks 1 to 4) minus the number of monthly migraine days during the OP.
Time Frame: OP and Weeks 1 to 4 of the DBT phase
Population: The analysis was performed on evaluable mITT participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: migraine days per month
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 348 | 347
migraine days per month | -2.9 [-3.32 to -2.46] | -1.7 [-2.15 to -1.29]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation in the DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition on-treatment in a patient or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. An SAE was defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received rimegepant; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
Time Frame: Weeks 1 to 12 of the DBT phase
Population: The analysis was performed on the participants treated in the DBT phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 370 | 371
Participants
  AEs | 133 | 133
  SAEs | 3 | 4
  AEs leading to study drug discontinuation | 7 | 4

7. Secondary Outcome: Number of Participants With AEs, SAEs, AEs Leading to Study Drug Discontinuation in the OLE Phase
Description: as for outcome 6
Time Frame: OLE Phase (Weeks 13 through 64)
Population: Open-Label (OL) rimegepant treated participants included enrolled participants who received at least one dose of OL rimegepant (non-missing OL rimegepant start date).
Measure: Count of Participants; unit: Participants
Groups:
- DBT Rimegepant/OL Rimegepant; DBT Placebo/OL Rimegepant: OLE Phase (Weeks 13 through 64): After completion of DBT phase, participants who continued to meet study entry criteria and had acceptable laboratory test results per protocol, entered the OLE phase and received a single oral dose of rimegepant 75 mg tablet EOD for 52 weeks. If participants had a migraine on a day that they were not scheduled to dose with rimegepant, they could take one tablet of rimegepant 75 mg on that calendar day to treat a migraine (PRN dosing).
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Number analyzed (Participants) | 302 | 301
Participants
  AEs | 150 | 162
  SAEs | 7 | 6
  AEs leading to study drug discontinuation | 9 | 8

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in the DBT Phase
Description: Clinically significant laboratory abnormalities were defined as Grade 3 to 4 laboratory test results according to numeric laboratory test criteria found in Common Technical Criteria for Adverse Events (CTCAE) Version 5.0 (2017) if available; otherwise, according to Division of Acquired Immune Deficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 (2017) for glucose, LDL-cholesterol, uric acid, and urinalysis. Laboratory test groups of clinical interest included hematology, serum chemistry, and urinalysis. Participants must have had a non-missing measurement in the DBT phase to be included for a given parameter.
Time Frame: Weeks 1 to 12 of the DBT phase
Population: The analysis was performed on the participants treated in the DBT phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 370 | 371
Participants
  Eosinophils: number analyzed (Participants) | 361 | 353
  Eosinophils | 0 | 0
  Hemoglobin: number analyzed (Participants) | 361 | 353
  Hemoglobin | 0 | 1
  Lymphocytes, high: number analyzed (Participants) | 361 | 353
  Lymphocytes, high | 0 | 0
  Lymphocytes, low: number analyzed (Participants) | 361 | 353
  Lymphocytes, low | 0 | 0
  Neutrophils: number analyzed (Participants) | 361 | 353
  Neutrophils | 4 | 2
  Platelets: number analyzed (Participants) | 360 | 353
  Platelets | 1 | 0
  White Blood Cells: number analyzed (Participants) | 361 | 353
  White Blood Cells | 1 | 0
  Alanine Aminotransferase (ALT): number analyzed (Participants) | 363 | 359
  Alanine Aminotransferase (ALT) | 1 | 0
  Aspartate Aminotransferase (AST): number analyzed (Participants) | 363 | 359
  Aspartate Aminotransferase (AST) | 1 | 0
  Albumin: number analyzed (Participants) | 361 | 354
  Albumin | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 363 | 359
  Alkaline Phosphatase | 0 | 0
  Bicarbonate: number analyzed (Participants) | 361 | 354
  Bicarbonate | 0 | 0
  Bilirubin: number analyzed (Participants) | 363 | 359
  Bilirubin | 0 | 0
  Calcium, high: number analyzed (Participants) | 361 | 354
  Calcium, high | 0 | 0
  Calcium, low: number analyzed (Participants) | 361 | 354
  Calcium, low | 0 | 0
  Cholesterol: number analyzed (Participants) | 43 | 57
  Cholesterol | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 361 | 354
  Creatine Kinase | 4 | 4
  Creatinine: number analyzed (Participants) | 361 | 354
  Creatinine | 0 | 0
  Glucose, high: number analyzed (Participants) | 360 | 354
  Glucose, high | 0 | 0
  Glucose, low: number analyzed (Participants) | 360 | 354
  Glucose, low | 0 | 0
  LDL-cholesterol: number analyzed (Participants) | 41 | 57
  LDL-cholesterol | 2 | 0
  LDL-cholesterol, fasting: number analyzed (Participants) | 18 | 26
  LDL-cholesterol, fasting | 0 | 0
  LDL-cholesterol, not fasting: number analyzed (Participants) | 23 | 31
  LDL-cholesterol, not fasting | 2 | 0
  Lactate Dehydrogenase: number analyzed (Participants) | 361 | 354
  Lactate Dehydrogenase | 0 | 0
  Potassium, high: number analyzed (Participants) | 361 | 354
  Potassium, high | 1 | 2
  Potassium, low: number analyzed (Participants) | 361 | 354
  Potassium, low | 0 | 0
  Sodium, high: number analyzed (Participants) | 361 | 354
  Sodium, high | 0 | 0
  Sodium, low: number analyzed (Participants) | 361 | 354
  Sodium, low | 0 | 0
  Triglycerides: number analyzed (Participants) | 43 | 57
  Triglycerides | 0 | 0
  Triglycerides, fasting: number analyzed (Participants) | 18 | 26
  Triglycerides, fasting | 0 | 0
  Triglycerides, not fasting: number analyzed (Participants) | 25 | 31
  Triglycerides, not fasting | 0 | 0
  Uric acid: number analyzed (Participants) | 361 | 354
  Uric acid | 0 | 0
  Glomerular Filtration Rate, Estimated: number analyzed (Participants) | 361 | 354
  Glomerular Filtration Rate, Estimated | 1 | 0
  Urine Glucose: number analyzed (Participants) | 49 | 55
  Urine Glucose | 0 | 0
  Urine Protein: number analyzed (Participants) | 46 | 55
  Urine Protein | 1 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in the OLE Phase
Description: Clinically significant laboratory abnormalities were defined as Grade 3 to 4 laboratory test results according to numeric laboratory test criteria found in CTCAE Version 5.0 (2017) if available; otherwise, according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 (2017) for glucose, LDL-cholesterol, uric acid, and urinalysis. Laboratory test groups of clinical interest included hematology, serum chemistry, and urinalysis. Participants must have had a non-missing measurement in the OLE phase to be included for a given parameter.
Time Frame: OLE Phase (Weeks 13 through 64)
Population: OL rimegepant treated participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Number analyzed (Participants) | 297 | 296
Participants
  Eosinophils: number analyzed (Participants) | 293 | 291
  Eosinophils | 0 | 0
  Hemoglobin: number analyzed (Participants) | 293 | 292
  Hemoglobin | 1 | 1
  Lymphocytes, high: number analyzed (Participants) | 293 | 292
  Lymphocytes, high | 0 | 0
  Lymphocytes, low: number analyzed (Participants) | 293 | 292
  Lymphocytes, low | 1 | 0
  Neutrophils: number analyzed (Participants) | 293 | 292
  Neutrophils | 1 | 1
  Platelets: number analyzed (Participants) | 293 | 292
  Platelets | 0 | 0
  White Blood Cells: number analyzed (Participants) | 293 | 292
  White Blood Cells | 0 | 0
  Alanine Aminotransferase (ALT) | 0 | 5
  Aspartate Aminotransferase (AST) | 1 | 3
  Albumin: number analyzed (Participants) | 294 | 292
  Albumin | 0 | 0
  Alkaline Phosphatase | 0 | 0
  Bicarbonate: number analyzed (Participants) | 294 | 292
  Bicarbonate | 0 | 0
  Bilirubin | 0 | 0
  Calcium, high: number analyzed (Participants) | 294 | 292
  Calcium, high | 0 | 0
  Calcium, low: number analyzed (Participants) | 294 | 292
  Calcium, low | 0 | 0
  Cholesterol: number analyzed (Participants) | 278 | 285
  Cholesterol | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 294 | 292
  Creatine Kinase | 4 | 7
  Creatinine: number analyzed (Participants) | 294 | 292
  Creatinine | 0 | 0
  Glucose, high: number analyzed (Participants) | 293 | 292
  Glucose, high | 0 | 0
  Glucose, low: number analyzed (Participants) | 293 | 292
  Glucose, low | 0 | 1
  LDL-cholesterol: number analyzed (Participants) | 275 | 283
  LDL-cholesterol | 5 | 5
  LDL-cholesterol, fasting: number analyzed (Participants) | 144 | 146
  LDL-cholesterol, fasting | 2 | 3
  LDL-cholesterol, not fasting: number analyzed (Participants) | 171 | 182
  LDL-cholesterol, not fasting | 3 | 2
  Lactate Dehydrogenase: number analyzed (Participants) | 294 | 292
  Lactate Dehydrogenase | 0 | 0
  Potassium, high: number analyzed (Participants) | 294 | 292
  Potassium, high | 2 | 0
  Potassium, low: number analyzed (Participants) | 294 | 292
  Potassium, low | 0 | 0
  Sodium, high: number analyzed (Participants) | 294 | 292
  Sodium, high | 0 | 0
  Sodium, low: number analyzed (Participants) | 294 | 292
  Sodium, low | 0 | 0
  Triglycerides: number analyzed (Participants) | 278 | 285
  Triglycerides | 3 | 2
  Triglycerides, fasting: number analyzed (Participants) | 144 | 148
  Triglycerides, fasting | 0 | 1
  Triglycerides, not fasting: number analyzed (Participants) | 174 | 183
  Triglycerides, not fasting | 3 | 2
  Uric acid: number analyzed (Participants) | 294 | 292
  Uric acid | 0 | 0
  Glomerular Filtration Rate, Estimated: number analyzed (Participants) | 294 | 292
  Glomerular Filtration Rate, Estimated | 0 | 0
  Urine Glucose: number analyzed (Participants) | 222 | 238
  Urine Glucose | 0 | 0
  Urine Protein: number analyzed (Participants) | 220 | 237
  Urine Protein | 0 | 0

10. Secondary Outcome: Number of Participants With Elevations of AST or ALT > 3 x Upper Limit of Normal (ULN) Concurrent With Total Bilirubin (TBL) > 2 x ULN During the DBT Phase
Description: Elevations of AST or ALT > 3 x ULN concurrent with TBL > 2 x ULN were defined as elevations on the same collection date. Participants must have had a non-missing AST, ALT, or TBL measurement in the OLE phase to be included.
Time Frame: Weeks 1 to 12 of the DBT phase
Population: The analysis was performed on the participants treated in the DBT phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 370 | 371
Percentage of participants | 0 [0.00 to 1.24] | 0 [0.00 to 1.24]

11. Secondary Outcome: Percentage of Participants With Elevations of AST or ALT > 3 x ULN Concurrent With TBL > 2 x ULN During the OLE Phase
Description: Elevations of AST or ALT > 3 x ULN concurrent with TBL > 2 x ULN were defined as elevations on the same collection date. Participants must have had a non-missing AST, ALT, or TBL measurement in the DBT phase to be included.
Time Frame: OLE Phase (Weeks 13 through 64)
Population: OL rimegepant treated participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Number analyzed (Participants) | 297 | 296
Percentage of participants | 0 [0.00 to 1.51] | 0 [0.00 to 1.52]

12. Secondary Outcome: Number of Participants With Hepatic-related AEs and Hepatic-related AEs Leading to Discontinuation During the DBT Phase
Description: Hepatic AEs were defined as all preferred terms in the DBT phase under the "Hepatic Disorders" Standardized Medical Dictionary (Version 21.1) for Regulatory Activities Query (SMQ), except those preferred terms in the "Congenital, Familial, Neonatal and Genetic Disorders of the Liver" SMQ.
Time Frame: Weeks 1 to 12 of the DBT phase
Population: The analysis was performed on the participants treated in the DBT phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 370 | 371
Participants
  Hepatic-related AE | 6 | 2
  Severe hepatic-related AE | 0 | 0
  Hepatic-related SAE | 0 | 0
  Hepatic-related AE leading to study drug discontinuation | 2 | 2

13. Secondary Outcome: Number of Participants With Hepatic-related AEs and Hepatic-related AEs Leading to Discontinuation During the OLE Phase
Description: Hepatic AEs were defined as all preferred terms in the OLE phase under the "Hepatic Disorders" SMQ, except those preferred terms in the "Congenital, Familial, Neonatal and Genetic Disorders of the Liver" SMQ.
Time Frame: OLE Phase (Weeks 13 through 64)
Population: OL rimegepant treated participants were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OL Rimegepant | DBT Placebo/OL Rimegepant
Number analyzed (Participants) | 302 | 301
Participants
  Hepatic-related AE | 2 | 9
  Severe hepatic-related AE | 0 | 1
  Hepatic-related SAE | 0 | 0
  Hepatic-related AE leading to study drug discontinuation | 1 | 1

14. Secondary Outcome: Mean Change From Baseline in the Migraine Specific Quality of Life (MSQoL) Role Function-Restrictive Domain Score at Week 12 of the DBT Phase
Description: The Migraine Specific Quality of Life (MSQoL) is a self-administered, 14-item instrument that has been validated in 3 domains: role restriction, role prevention, and the emotional function. The role function-restrictive domain consists of 7 items that describe how migraine limits one's daily social and work-related activities. Participants respond to items using a 6-point scale: "none of the time," "a little bit of the time," "some of the time," "a good bit of the time," "most of the time," and "all of the time," which are assigned scores of 1 to 6, respectively. Item scores are recoded using (7 - original score). Next, raw dimension scores are computed as a sum of recoded item scores and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life.
  The change from baseline was calculated as the MSQoL restrictive role function domain score at Week 12 of the DBT phase minus the MSQoL restrictive role function domain score at baseline.
Time Frame: Baseline, Week 12 of the DBT Phase
Population: The analysis was performed on evaluable mITT participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 269 | 266
score on a scale | 18.0 [15.54 to 20.56] | 14.6 [12.07 to 17.10]

15. Secondary Outcome: Mean Change From Baseline in the Migraine Disability Assessment (MIDAS) Total Score at Week 12 of the DBT Phase
Description: The Migraine Disability Assessment (MIDAS) is a retrospective, self-administered, 5-item questionnaire that measures headache-related disability as lost time due to headache from paid work or school, household work, and non-work activities. Participants provide the number of missed work or school days; missed household chores days; missed social or leisure activity days; and days at work or school, and separately at home, where productivity was reduced by half or more in the last 3 months (scale: 0 - 90 for each of 5 subscales). The 5 subscale scores are summed to compute the MIDAS total score (scale: 0 - 450). Lower scores indicate less headache-related disability.
  The change from baseline was calculated as the MIDAS total score at Week 12 of the DBT phase minus the MIDAS total score at baseline.
Time Frame: Baseline, Week 12 of the DBT Phase
Population: The analysis was performed on evaluable mITT participants
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 269 | 266
Scores on a scale | -11.8 [-15.41 to -8.21] | -11.7 [-15.29 to -8.10]

ADVERSE EVENTS:
Time Frame: DBT Phase: From the first dose in the DBT Phase (Week 1) to Week 12 OLE Phase: Week 13 to Week 64 Follow-up phase: 8 weeks after the end of treatment (maximum duration of treatment: 64 weeks)
Description: AEs are presented according to the periods of the study.
  Randomized phase: Participants treated in the DBT phase were included.
  OLE phase: OL rimegepant treated participants included enrolled participants who received at least one dose of OL rimegepant (non-missing OL rimegepant start date).
  Follow-up phase: Follow-up participants included all treated participants whose last contact date was in the follow-up safety analysis period.
Groups:
- DBT Rimegepant/OLE Rimegepant - OLE Phase: OLE Phase (Weeks 13 through 64): After completion of DBT phase, participants, who continued to meet study entry criteria and had acceptable laboratory test results per protocol, entered the OLE phase and received a single oral dose of rimegepant 75 mg tablet EOD for 52 weeks. If participants had a migraine on a day that they were not scheduled to dose with rimegepant, they could take one tablet of rimegepant 75 mg on that calendar day to treat a migraine (as needed [PRN] dosing).
- DBT Placebo/OLE Rimegepant - OLE Phase: OLE Phase (Weeks 13 through 64): After completion of DBT phase, participants, who continued to meet study entry criteria and had acceptable laboratory test results per protocol, entered the OLE phase and received a single oral dose of rimegepant 75 mg tablet EOD for 52 weeks. If participants had a migraine on a day that they were not scheduled to dose with rimegepant, they could take one tablet of rimegepant 75 mg on that calendar day to treat a migraine (PRN dosing).
- DBT Rimegepant/OLE Rimegepant - Follow-up Phase: Participants received rimegepant during the DBT phase (Week 1 to Week 12) and OLE phase (Week 13 to Week 64). After completing the OLE phase, participants had follow-up safety visits 2 and 8 weeks after the EOT visit. Participants who did not complete the DBT phase and/or did not enter or complete the OLE phase were to complete the EOT visit, the 2-week follow-up safety visit, and the 8-week follow-up safety visit after their early discontinuation.
- DBT Placebo/OLE Rimegepant - Follow-up Phase: Participants received placebo during the DBT phase (Week 1 to Week 12) and rimegepant OLE phase (Week 13 to Week 64). After completing the OLE phase, participants had follow-up safety visits 2 and 8 weeks after the EOT visit. Participants who did not complete the DBT phase and/or did not enter or complete the OLE phase were to complete the EOT visit, the 2-week follow-up safety visit, and the 8-week follow-up safety visit after their early discontinuation.
Arm/Group | Rimegepant - Randomization Phase | Placebo - Randomization Phase | DBT Rimegepant/OLE Rimegepant - OLE Phase | DBT Placebo/OLE Rimegepant - OLE Phase | DBT Rimegepant/OLE Rimegepant - Follow-up Phase | DBT Placebo/OLE Rimegepant - Follow-up Phase
All-Cause Mortality (participants affected / at risk) | 0/370 | 0/371 | 1/302 | 1/301 | 0/332 | 0/336
Serious Adverse Events (participants affected / at risk) | 3/370 | 4/371 | 7/302 | 6/301 | 2/332 | 2/336
Other Adverse Events (participants affected / at risk) | 0/370 | 0/371 | 41/302 | 37/301 | 41/332 | 34/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant - Randomization Phase (N=370) | Placebo - Randomization Phase (N=371) | DBT Rimegepant/OLE Rimegepant - OLE Phase (N=302) | DBT Placebo/OLE Rimegepant - OLE Phase (N=301) | DBT Rimegepant/OLE Rimegepant - Follow-up Phase (N=332) | DBT Placebo/OLE Rimegepant - Follow-up Phase (N=336)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depressive delusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant - Randomization Phase (N=370) | Placebo - Randomization Phase (N=371) | DBT Rimegepant/OLE Rimegepant - OLE Phase (N=302) | DBT Placebo/OLE Rimegepant - OLE Phase (N=301) | DBT Rimegepant/OLE Rimegepant - Follow-up Phase (N=332) | DBT Placebo/OLE Rimegepant - Follow-up Phase (N=336)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 21 | 22 | 21 | 19
Nasopharyngitis (Infections and infestations) | 0 | 0 | 23 | 15 | 23 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is less than or equal to 60 days from the date that the communication is submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03732638/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03732638/SAP_002.pdf